CLINICAL TRIAL: NCT01012908
Title: Clinical Non-Inferiority of Pancreatic Enzymes (Norzyme ® - Bergamo) Compared To Creon ® (Solvay Pharmaceutical) in Patients With Exocrine Pancreatic Insufficiency
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Azidus Brasil (Industry)
Responsible Party: Alexandre Frederico, LAL Clinica Pesquisa e Desenvolvimento Ltda
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PANBER0609
Record Dates: First submitted 2009-11-11; First posted 2009-11-13 (Estimated); Last update posted 2010-10-28 (Estimated); Status verified 2009-11

CONDITIONS: Pancreatic Insufficiency
MeSH Terms: conditions — Exocrine Pancreatic Insufficiency | interventions — Pancrelipase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Norzyme (Experimental): Pancreatic Enzymes - Norzyme (Bergamo)
  Interventions: Dietary Supplement: Norzyme - Bergamo
- Creon (Solvay) (Active Comparator): Pancreatic Enzymes - Creon (Solvay)
  Interventions: Dietary Supplement: Creon

INTERVENTIONS:
Dietary Supplement: Norzyme - Bergamo — 2 - 8 tablets per day.
  Arms: Norzyme
Dietary Supplement: Creon — 2 - 8 tablets pet day
  Arms: Creon (Solvay)

SUMMARY:
The primary objective of this clinical trial is to demonstrate non-inferiority clinical development of pancreatic enzymes from Laboratory Bergamo (Norzyme ®) in relation to pancreatic enzymes from Solvay Pharmaceuticals (Creon ®), by comparing the average amount of lipids in the feces of 72 hours after 14 days of treatment with each drug.

DETAILED DESCRIPTION:
As a secondary objective will be assessed the following parameters:

* Incidence of abdominal pain;
* Frequency of flatus;
* Frequency of bowel movements during the treatment;
* Consistency of stools during treatment;
* Amount of medication used among the treatments. All these parameters will be measured based on reports of patients in a specific diary.

ELIGIBILITY:
Inclusion Criteria:

* Patients must agree with the purposes of the study and sign the Informed Consent in two ways;
* Be aged over 18 years;
* Display chronic exocrine pancreatic insufficiency due to chronic pancreatic, post surgical or other situation that leads to severe glandular disease;
* Doing controlled clinical treatment of enzyme replacement with Creon ® 25,000 (or similar with the same concentration of lipase) during meals;
* Agree to record daily food intake in phase 2 and repeat the diet in phase 3;
* Present ability to meet the patient's diary;
* Be clinically compensated with replacement therapy;
* Must be admitted patients in both the sexes;
* Must be accepted patients of any ethnicity.

Exclusion Criteria:

* Cystic fibrosis;
* Acute pancreatitis;
* Participation in any experimental study or ingestion of any experimental drug in the 12 months preceding the study;
* Diabetes decompensated;
* Regular use of medications that interfere with the action of the drug test: the 4 weeks preceding the study or any medication that interferes with the drug test a week before the start of the study;
* Any type of treatment for morbid obesity;
* Abusive use of alcohol in the three months preceding the study;
* Pregnancy and lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2010-03; Primary Completion 2010-04 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Amount of fat in the stools of 72 hours of medication use between the two treatments. | First period: 12th, 13th and14th day. Second period (After crossover medication): 12th, 13th and14th day

SECONDARY OUTCOMES:
Frequency of bowel movements per day | First period: days 1 - 14. Second period: days 1-14. (every day)
Consistency and characteristics of feces | First period: days 1 - 14. Second period: days 1-14. (every day)
Frequency and intensity of abdominal pain daily | First period: days 1 - 14. Second period: days 1-14. (every day)
Frequency of flatulence daily | First period: days 1 - 14. Second period: days 1-14. (every day)
Amount of drug used in treatment | First period: days 1 - 14. Second period: days 1-14. (every day)

CONTACTS AND LOCATIONS:
Locations (1):
- Lal Clinica Pesquisa E Desenvolvimento Ltda, Valinhos, São Paulo, Brazil